CLINICAL TRIAL: NCT05549115
Title: Susceptibility-Guided Sequential Therapy Versus Empirical Therapy for Helicobacter Pylori Infection: a Randomised Controlled Trial
Brief Title: Susceptibility-Guided Sequential Therapy for Helicobacter Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liaocheng People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS-HP001
Record Dates: First submitted 2022-09-18; First posted 2022-09-22 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2022-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Drug Resistance, Microbial; Microbial Sensitivity Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- clarithromycin-sensitive(first-line) (Experimental): If H. pylori is sensitive to clarithromycin, we will administer clarithromycin triple therapy-esomeprazole (20 mg, twice daily), clarithromycin (500 mg, twice daily), and amoxicillin (1.0 g, twice daily)-for 14 days
  Interventions: Drug: clarithromycin-sensitive(first-line)
- clarithromycin-resistant(first-line) (Experimental): If H. pylori is clarithromycin resistance, we selected the High-dose dual therapy (HDDT) regimen as first-line treatment. HDDT-esomeprazole (20 mg, four times daily) and amoxicillin (750 mg, four times daily)-will be used for 14 days.
  Interventions: Drug: clarithromycin-resistant(first-line)
- empirical therapy group first-line (Active Comparator): The empirical therapy group will receive Bismuth-containing quadruple therapy(BQT) as first-line treatment, The BQT regime is comprising of esomeprazole (20 mg, twice daily), colloidal bismuth pectin (150 mg, four times daily), clarithromycin (500 mg, twice daily), and amoxicillin (1.0 g, twice daily) for 14 days.
  Interventions: Drug: empirical therapy group first-line
- levofloxacin-sensitive(rescue treatment) (Experimental): If H. pylori was levofloxacin-sensitive, we will use the levofloxacin quadruple regimen as rescue treatment-esomeprazole (20 mg, twice daily), levofloxacin (500 mg, once daily), amoxicillin (1.0 g, twice daily), and colloidal bismuth pectin (150 mg, four times daily)-for 14 days.
  Interventions: Drug: levofloxacin-sensitive(rescue treatment)
- levofloxacin-resistant(rescue treatment) (Experimental): If H. pylori was levofloxacin-resistant, we will use furazolidone quadruple regimen as rescue treatment-esomeprazole (20 mg, twice daily), furazolidone (100 mg, twice daily), amoxicillin (1.0 g, twice daily), and colloidal bismuth pectin (150 mg, four times daily)-for 14 days.
  Interventions: Drug: levofloxacin-resistant(rescue treatment)
- empirical therapy group rescue treatment (Active Comparator): If BQT fails, HDDT-esomeprazole (20 mg, four times daily) and amoxicillin (750 mg, four times daily)-will be used as a rescue treatment for 14 days.
  Interventions: Drug: empirical therapy group rescue treatment

INTERVENTIONS:
Drug: clarithromycin-sensitive(first-line) — esomeprazole (20 mg, twice daily), clarithromycin (500 mg, twice daily), and amoxicillin (1.0 g, twice daily) for 14 days
  Other Names: clarithromycin triple therapy
  Arms: clarithromycin-sensitive(first-line)
Drug: clarithromycin-resistant(first-line) — esomeprazole (20 mg, four times daily) and amoxicillin (750 mg, four times daily) for 14 days
  Other Names: High-dose PPI-amoxicillin dual therapy
  Arms: clarithromycin-resistant(first-line)
Drug: empirical therapy group first-line — esomeprazole (20 mg, twice daily), colloidal bismuth pectin (150 mg, four times daily), clarithromycin (500 mg, twice daily), and amoxicillin (1.0 g, twice daily) for 14 days
  Other Names: Bismuth-containing quadruple therapy
  Arms: empirical therapy group first-line
Drug: levofloxacin-sensitive(rescue treatment) — esomeprazole (20 mg, twice daily), levofloxacin (500 mg, once daily), amoxicillin (1.0 g, twice daily), and colloidal bismuth pectin (150 mg, four times daily) for 14 days
  Other Names: levofloxacin quadruple regimen
  Arms: levofloxacin-sensitive(rescue treatment)
Drug: levofloxacin-resistant(rescue treatment) — esomeprazole (20 mg, twice daily), furazolidone (100 mg, twice daily), amoxicillin (1.0 g, twice daily), and colloidal bismuth pectin (150 mg, four times daily) for 14 days
  Other Names: furazolidone quadruple regimen
  Arms: levofloxacin-resistant(rescue treatment)
Drug: empirical therapy group rescue treatment — esomeprazole (20 mg, four times daily) and amoxicillin (750 mg, four times daily) for 14 days
  Other Names: High-dose PPI-amoxicillin dual therapy
  Arms: empirical therapy group rescue treatment

SUMMARY:
The main objective of this trial is to assess whether a sequential therapy strategy based on molecular antibiotic susceptibility testing (including clarithromycin and fluoroquinolone) for H. pylori infection will improve the eradication rate compared to an empirical therapy.

DETAILED DESCRIPTION:
This trial is designed as a prospective, randomised, open-label, active-controlled and single-centre study. For empirical therapy group(control group), Bismuth quadruple therapy will be an empirical first-line therapy, and high dose dual (proton-pump inhibitor + amoxicillin) treatment will be for rescue therapy if the first-line empirical treat failure. For the susceptibility-guided sequential therapy group, regimens were selected based on H. pylori susceptibility to clarithromycin and levofloxacin. The primary outcome is the first-line eradication rate in both groups, and the overall (including first- and rescue therapies) H. pylori eradication rates in both groups is one of the secondary outcomes. The eradication rates of H. pylori will be analysed by intention-to-treat analysis, modified intention-to-treat analysis and per-protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori infection was determined using at least one of the following tests: 13C/14C-urea breath test (UBT), stool H. pylori antigen test, rapid urease test, and histological analysis within 4 weeks.
* Patients were naïve to H. pylori treatment.

Exclusion Criteria:

* Allergy to any drug administered.
* Pregnancy and lactation.
* Major systemic diseases, such as severe cardiopulmonary or liver dysfunction.
* Complicated with active peptic ulcer disease, gastric cancer, or prior gastrectomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
the first-line H. pylori eradication rate | 4-8 weeks after the end of treatment.
  the proportion of participants with successful H. pylori eradication, as determined by 13C-Urea breath test(UBT), at least 4 weeks after the end of the first-line treatment period between Susceptibility-guided therapy(SGT) and empirical therapy(ET) group.

SECONDARY OUTCOMES:
the rescue H. pylori eradication rate | 4-8 weeks after the second treatment
  The second line eradication rate between SGT and ET group.
the overall H.pylori eradication rate | 4-8 weeks after the second treatment
  the total H.pylori eradication rate (first-line and second-line)between SGT and ET group.
high-dose dual therapy eradication rate | 4-8 weeks after the second treatment
  compare H. pylori eradication rate between clarithromycin resistance group and empirical BQT failure group.
Adverse events and compliance | 3 days after the end of treatment.
  3 days after the completion of therapy according to a data collection form

CONTACTS AND LOCATIONS:
Overall Officials: Jing run Zhao, Dr, Study Chair — Liaocheng People's Hospital
Locations (1):
- Liaocheng people's hospital, Liaocheng, Shandong, China

REFERENCES:
- [Derived] Lu K, Lang C, Zou X, Zang L, Sang W, Feng Q, Mu Y, Liu L, Xu C, Zhao J. Susceptibility-guided sequential strategy versus empirical therapy for Helicobacter pylori infection: study protocol for a randomised controlled trial. Trials. 2023 Jun 19;24(1):413. doi: 10.1186/s13063-023-07457-z. PMID 37337241